CLINICAL TRIAL: NCT06834100
Title: Simple Blinded Multicenter Randomized Comparative Study to Assess Immunogenicity, Reactogenicity and Safety of the Drug GNG-DE
Brief Title: Assessment of Immunogenicity, Reactogenicity and Safety of the Drug GNG-DE in Comparison With the Reference Drug
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: NPO Petrovax (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: GNG-DE-III-24
Record Dates: First submitted 2025-02-13; First posted 2025-02-19 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-11

CONDITIONS: Infections; Meningococcal
MeSH Terms: conditions — Infections

STUDY DESIGN:
Intervention Model Description: In the study, 240 subjects aged 3-55 years (inclusive) meeting the eligibility criteria and not meeting any non-eligibility criteria will be randomized, of which there are 80 adult volunteers aged 18-55 years inclusive, 80 adolescents aged 11-17 years inclusive, 80 children aged 3-10 years inclusive. Taking into account the possible withdrawal at the screening stage, the maximum number of subjects included in the study will be no more than 260.
Who Masked: Participant
Masking Description: The subject will be randomly assigned (using a computer program) to one of two groups:
  The 1st group (n=40) of participants will receive the drug GNG-DE in a dose of 0.5 ml intramuscularly into the deltoid muscle area.
  The 2nd group (n=40) of participants will receive Menactra® in a dose of 0.5 ml intramuscularly into the deltoid muscle area.
  This study will be conducted as a single blind study, i.e. The study physician will know, but the subject will not know, which drug (study or reference drug) will be administered.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Stage I (Experimental): At this stage, adult volunteers aged 18-55 years old (inclusive) will be enrolled in the study. After screening procedures, 80 volunteers who meet the eligibility criteria and do not meet any non-eligibility criteria will be randomized into 2 groups in a 1: 1 ratio
  Interventions: Drug: polysaccharide conjugated vaccine for prevention of meningococcal infection of serogroups A, C, W, Y
- Stage II (Experimental): Stage II will begin after receiving the positive conclusion of the IDMC on the basis of the consideration of stage I data. At this stage, adolescents aged 11-17 years old (inclusive) will be included in the study. After screening procedures, 80 adolescents who meet the eligibility criteria and do not meet any non-eligibility criteria will be randomized into 2 groups in a 1:1 ratio
  Interventions: Drug: polysaccharide conjugated vaccine for prevention of meningococcal infection of serogroups A, C, W, Y
- Stage III (Experimental): Stage III will begin after receiving the positive conclusion of the IDMC on the basis of the consideration of stage II data. At this stage, children aged 3-10 years old (inclusive) will be included in the study. After screening procedures, 80 children who meet the eligibility criteria and do not meet any non-eligibility criteria will be randomized into 2 groups in a 1:1 ratiowill receive Menactra® at a dose of 0.5 mL intramuscularly into the deltoid site.
  Interventions: Drug: polysaccharide conjugated vaccine for prevention of meningococcal infection of serogroups A, C, W, Y

INTERVENTIONS:
Drug: polysaccharide conjugated vaccine for prevention of meningococcal infection of serogroups A, C, W, Y — Group 1 (n = 40) will receive GNG-DE at a dose of 0.5 mL intramuscularly into the deltoid site.
  Group 2 (n = 40) will receive Menactra® at a dose of 0.5 mL intramuscularly into the deltoid site.

SUMMARY:
Assessment of immunogenicity, reactogenicity and safety of GNG-DE in comparison with the reference drug

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects aged 3-55 years old inclusive at the time of screening beginning.
2. Availability of a signed Volunteer Informed Consent Form (Volunteer Information Sheet, VIS) (for participants aged 7-55 years inclusive) and/or the parent/adoptive parent informed consent form (Parent Information Sheet, PIS) signed by one of parents/adoptive parents (for participants aged 3-17 years old inclusive).
3. Negative result of SARS-CoV-2 antigen rapid test at screening.
4. Negative pregnancy test result in fertile females of reproductive age. For females not reached puberty, and for girls/women unable to childbirth (with past infertility, hysterectomy, bilateral oophorectomy, bilateral tubal ligation, menopause for more than 2 years), the pregnancy test shall not be performed.
5. For participants of 14-55 years old inclusive with preserved reproductive function, the consent to use of reliable methods of contraception (abstinence, condoms in combination with spermicide and/or hormonal contraception) during the study.

   For participants aged 3-13 years old inclusive and females incapable of childbearing, the consent to use reliable methods of contraception is not required.
6. The consent of a participant and/or a parent/an adoptive parent of a participant to cooperate in good faith with the investigator and the center staff, come to appointed visits, fill out the observation diary and comply with the requirements of the Protocol.

Exclusion Criteria:

1. Hypersensitivity to any component of the test/reference drug.
2. Evident severe systemic reactions to any vaccines in anamnesis.
3. Impossibility of intramuscular injections.
4. Changes in the skin (pigmentation, tattoo, scars etc.) at the planned injection site of the test/reference drug (the deltoid muscle area).
5. Acute infectious and non-infectious diseases, exacerbation of chronic diseases at screening or less than 14 days before screening.
6. Body temperature measured in the armpit ≥ 37.0°C at Visits 0 and 1.
7. The history of chronic diseases that are significant in the opinion of the investigator (for example, malignant neoplasms, blood diseases, autoimmune diseases, immunodeficiencies, etc.).
8. The history of meningococcal infection.
9. Contact with a person with the confirmed infection caused by N. meningitidis less than 2 months before screening.
10. The history of convulsive syndrome or the advanced neurological disease.
11. The history of Guillain-Barré syndrome.
12. The history of mental diseases.
13. Drug administration:

    * the history of meningococcal mono- or polyvalent vaccine, influenza vaccine within 14 days before screening, other vaccines within 30 days before screening;
    * immunostimulants less than 30 days before screening;
    * the immunosuppressive therapy, including systemic corticosteroids, prescribed for more than 5 days, or in the daily dose of more than 1 mg/kg/day of prednisolone or its equivalent - less than 30 days before screening;
    * antipyretics, analgesics - for less than 24 hours before Visits 0 and 1;
    * systemic antibacterial drugs-- for less than 72 hours before Visits 0 and 1;
    * anticoagulants - for less than 3 weeks before Visits 0 and 1;
    * immunoglobulins, blood or plasma products - for less than 3 months before Visits 0 and 1.
14. Planning the administration of vaccines with the exception of the test/reference drug during the clinical study.
15. Surgical interventions performed less than 3 months before screening.
16. Participation in another clinical study less than 30 days before screening.
17. Other conditions that, in the opinion of the investigator, interfere to the enrollment.

Ages: 3 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-02-12 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary immunogenicity parameter | Day 29 ± 1
  Proportion (frequency) of subjects with seroconversion to meningococcal serogroups A, C, Y and W135 Seroconversion is defined as (for each serogroup it is determined separately)

SECONDARY OUTCOMES:
Secondary immunogenicity parameters | Day 29 ± 1
  The proportion (frequency) of vaccinated subjects with seroprotection
Secondary immunogenicity parameters | Day 29 ± 1
  Geometric mean titers of SBA to antigens of meningococcal serogroups A, C, Y and W135

OTHER OUTCOMES:
SAFETY ASSESSMENT | 1-7 days after vaccination, including the day of vaccination
  Criteria for assessing reactogenicity :
  * The proportion (frequency) of vaccinated subjects with expected local reactions (pain, redness, swelling) of any severity.
  * The proportion (frequency) of vaccinated subjects with expected systemic reactions (fever (according to measurement of body temperature in the armpit), gastrointestinal symptoms (abdominal pain, nausea, vomiting or diarrhea), headache, drowsiness, irritability, loss of appetite, arthralgia) of any severity.
  * The proportion (frequency) of vaccinated subjects with severe local reactions (pain, redness, swelling).
  * The proportion (frequency) of vaccinated subjects with severe systemic reactions (fever (according to measurement of body temperature in the armpit), gastrointestinal symptoms (abdominal pain, nausea, vomiting or diarrhea), headache, drowsiness, irritability, loss of appetite, arthralgia).

CONTACTS AND LOCATIONS:
Locations (16):
- Russia (16):
  - Federal State Budgetary Educational Institution of Higher Education "Kirov State Medical University" of the Ministry of Health of the Russian Federation, Kirov
  - Federal Budgetary Scientific Institution "Central Research Institute of Epidemiology" of the Federal Service for Surveillance on Consumer Rights Protection and Human Wellbeing, Moscow
  - Federal State Budgetary Scientific Institution "I.I. Mechnikov Research Institute of Vaccines and Serums", Moscow
  - Federal State Budgetary Scientific Institution "Russian Scientific Center of Surgery named after Academician B.V. Petrovsky", Moscow
  - State Budgetary Institution of Healthcare of the City of Moscow "Morozovskaya Children's City Clinical Hospital of the Moscow City Healthcare Department", Moscow
  - Federal State Budgetary Educational Institution of Higher Education "Perm State Medical University named after Academician E.A. Wagner" of the Ministry of Health of the Russian Federation, Perm
  - State Budgetary Healthcare Institution of Perm Krai "City Children's Clinical Polyclinic No. 5", Perm
  - Federal State Budgetary Institution "A. A. Smorodintsev Research Institute of Influenza" of the Ministry of Health of the Russian Federation, Saint Petersburg
  - Federal State Budgetary Institution "Children's Scientific and Clinical Center for Infectious Diseases of the Federal Medical and Biological Agency", Saint Petersburg
  - Limited Liability Company "Energy of Health", Saint Petersburg
  - Limited Liability Company "PiterClinic", Saint Petersburg
  - Saint Petersburg State Budgetary Healthcare Institution "Children's City Polyclinic No. 44", Saint Petersburg
  - Federal State Budgetary Educational Institution of Higher Education "National Research Mordovian State University named after N.P. Ogarev", Saransk
  - Limited Liability Company "DNA Research Center", Saratov
  - Federal State Budgetary Educational Institution of Higher Education "Smolensk State Medical University" of the Ministry of Health of the Russian Federation, Smolensk
  - State Budgetary Healthcare Institution of the Sverdlovsk Region "Central City Hospital No. 7, Yekaterinburg", Yekaterinburg